CLINICAL TRIAL: NCT03832101
Title: Improvement of Facial Recognition Ability and Multitasking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Christopher L. Asplund, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S-17-180
Record Dates: First submitted 2019-02-02; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Facial Discrimination; Multitasking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Difficult face discrimination (Experimental): All participants will complete 5 training and testing sessions in total, once a day, over the course of a week (weekdays). On the first day, participants will go through an initial test (Cambridge Face Memory Test; approximately 15 minutes) to determine their baseline facial recognition ability. Thereafter, participants in the Difficult group will undergo training involving discriminations between highly similar faces. Each participant's involvement in the study will last only 5 consecutive days. The total participation time is 7.5 hours per participant.
  Interventions: Behavioral: MATB
- Easy face discrimination (Experimental): All participants will complete 5 training and testing sessions in total, once a day, over the course of a week (weekdays). On the first day, participants will go through an initial test (Cambridge Face Memory Test; approximately 15 minutes) to determine their baseline facial recognition ability. Those in the Easy group will discriminate between dissimilar faces. Each participant's involvement in the study will last only 5 consecutive days. The total participation time is 7.5 hours per participant.
  Interventions: Behavioral: MATB
- Control (Active Comparator): All participants will complete 5 training and testing sessions in total, once a day, over the course of a week (weekdays). On the first day, participants will go through an initial test (Cambridge Face Memory Test; approximately 15 minutes) to determine their baseline facial recognition ability. Those in the Control group will perform a simple face-matching exercise. This training will last for approximately 30 minutes. Each participant's involvement in the study will last only 5 consecutive days. The total participation time is 7.5 hours per participant.
  Interventions: Behavioral: MATB

INTERVENTIONS:
Behavioral: MATB — MATB has two multitasking tasks and two attention tasks. The two multitasking tasks evaluates performance on multiple cognitively demanding assignments in both the auditory and visual domains. The two attention tasks measures performance in sustained and selective attention

SUMMARY:
This study aims to determine the efficacy of training on facial recognition and multitasking. The researchers hypothesize that participants who have undergone facial recognition and multitasking training will demonstrate an improved facial recognition ability and performance in multi-tasking. The researchers also hypothesize that measures of sustained and selective attention will predict performance on multitasking tasks. This work sets the ground work for future research into if and how facial recognition and multitasking ability can be improved.

DETAILED DESCRIPTION:
There has been evidence showing improvements on performance on various cognitive tasks after training, but evidence on multitasking and facial recognition is lacking. Both multi-tasking and facial recognition are crucial for military and law enforcement personnel, and the respective organizations can consider these abilities during their respective recruitment and training processes.

This study will test whether training on multi-tasking and facial recognition tasks can improve an individual's performance. Additionally, it will test whether their performance on other measures of attention and multitasking can predict changes post-training.

Participants will go through 5 testing sessions span over 5 days. For each session, participants will complete a multitasking task and a facial recognition task. Participants are hypothesized to improve in their performance after 5 consecutive days of training on these 2 tasks. Additionally, participants will also complete 2 attention tasks, 1 face memory task, and 1 other multi-tasking task only on the first day. Both multitasking tasks are expected to correlate at baseline, and performance on the attention tasks may predict performance on multitasking tasks as these tasks require sustained and selective attention. A face memory task will also be used to account for each individual's baseline facial recognition ability.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 21 if they are not from NUS or Yale-NUS. NUS or Yale-NUS students over 18 can also participate. All participants are expected to be fluent in English.

Exclusion Criteria:

* Participants with a history of perceptual or memory deficit will be excluded.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Facial recognition performance change during training | Day 1, 2, 3, 4, 5
  The crucial measure is percent correct recognition of target faces learned on the first day. These faces are either presented in isolation (Is this a target face? Yes/No) or with other faces (Which is the target?). Performance is measured on each day of training to establish learning trajectories.
Multi-tasking performance change during training | Day 1, 2, 3, 4, 5
  The crucial measures are speed and accuracy on each component task of the MATB (Multi-Attribute Task Battery; Comstock & Arnegard, 1992). Performance is measured on each day of training to establish learning trajectories.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided